CLINICAL TRIAL: NCT06591988
Title: A Multicenter Study to Identify Determinants Associated With Black Carbon Concentration in Biological Samples and Predictors of Quality of Life in Different Subpopulations Distinguished by Age Group and Residence
Brief Title: Environmental Pollutants and Life Quality
Acronym: ZEPHYR
Status: Enrolling by invitation | Type: Observational
Sponsor: Azienda Sanitaria Locale di Taranto (Other Government)
Responsible Party: Principal Investigator, Roberta Zupo, Principal Investigator, Azienda Sanitaria Locale di Taranto
Other Study IDs: 01/2024
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Environment; Pollution Exposure; Mortality; Healthcare; Lifestyle Factors
Keywords: environmental pollutants; lifestyle; mortality; risk factors; public health; life expectancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle factors — introduction of environmental risk mitigation policies, from data and evidence from case studies (several European cities) with different levels of exposure to environmental, health, geographic, and socioeconomic factors.
  Other Names: environmental risk mitigation policies

SUMMARY:
This study is part of the MISTRAL project, funded by the European Commission under the Horizon Europe Program, within the Work Programme 2021-2022 of Pillar II - Health Cluster on Environment and Health, which has the main objective of creating a cloud-based informatics platform for Health Impact Assessment analysis that, thanks to artificial intelligence, is able to simulate different clinical scenarios, economic and social, before and after the introduction of environmental risk mitigation policies, starting from data and evidence derived from case studies (several European cities) with different levels of exposure to environmental, health, geographical and socio-economic factors. The Project involves 11 partners distributed among Italy (Istituto Superiore di Sanità, Azienda Sanitaria Locale di Taranto, University of Bari, Politecnico di Bari, APS PLANET), Belgium (University of Hasselt), Poland (AGH-University of Technology and Science), Germany (Nuromedia), Spain (Ubitel), Greece (WINGS-ICT Solutions) and England (University of Oxford, University of Suffolk).

Specifically, the ZEPHYR study is a cross-sectional (cross-sectional), population-based, multicenter survey. The centers involved are the ASL of Taranto with the Taranto City Single District (Coordinating Recruitment Center), the University of Hasselt, Belgium (Recruitment Center Hasselt Hospital Campus), and the University of Krakow, Poland (Rybnik University Hospital as recruitment center).

DETAILED DESCRIPTION:
The purpose of the cross-sectional interventional survey is to directly measure the population most susceptible to environmental determinants, the frequency of multidimensional variables, and the conditions that may change their health status. Specifically, the survey has two main objectives, corresponding to two outcomes to be investigated separately in the same populations.

1. Recruitment of 380 children, 418 adults and 418 elderly. These sample sizes will be those planned for each unit (Taranto in Italy, Rybnik in Poland, and Genk-Hasselt County in Belgium).
2. The areas of Tamburi (an area presumably highly exposed to environmental pollutants) and Talsano-Lama-San Vito will be selected for sampling in the city of Taranto.
3. Administration of informed consents through general practitioners and pediatricians of free choice in the areas involved in recruitment.
4. Collection of urine and blood samples to measure determinants associated with the concentration of black carbon (BC) in urine samples and other pollutants (PCBs, Benzene) in blood and urine. The collected exposure data will be used to create a pragmatic score (dose-response function) of environmental pollution contamination.
5. Measurement of clinical, social and environmental determinants and predictors of quality of life (QoL), measured using a specific validated multinational questionnaire the EQ-5D-5L, and to create a probabilistic score, using feature selection algorithms in machine learning, that can predict different classes of QoL using clinical, social and environmental determinants.

Black carbon assay will be considered as a proxy for exposure to pollutants specifically related to steel production. This has been identified as one of the most promising biomarkers in terms of evidence of both deterministic and stochastic biological damage, in particular in the pediatric population,3 and it has even been demonstrated in fetal exposure4. In addition, the huge amount of urine samples collected will lead to the creation of a urine biobank for further (eventual) molecular analysis. Quality of life will be measured directly in different subpopulations, to be used to construct individual surrogate QALY scores.

On the sidelines of these macro objectives, however, additional biomarkers will be analyzed in the tissues of consenting subjects.

Specifically, the following will be analyzed :

1. Benzene metabolites: S-phenyl-mercapturic acid (SPMA)c,t- muconic acids;
2. metabolites of PAHs: the 1-hydroxypyrene (1-OHPyr)
3. cotinine to identify smokers, those exposed to secondhand smoke, and in nonsmokers.
4. PCR analysis for detection of telomere length (indicators of aging)

ELIGIBILITY:
Inclusion Criteria:

* Within the population of Taranto (southern Italy), healthy volunteer subjects will be recruited, and sampled from the following geographic areas of the city: the Tamburi district (an area presumably highly exposed to environmental pollutants), and the Talsano-Lama-San Vito district.

Exclusion Criteria:

* unhealthy subjects
* Taranto people residing outside the above areas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sampling frame will consist of the demographic dataset from regional health registries for each national unit. The survey will include children, adults, and the elderly, and probability sampling will be applied in each subpopulation, using a nearest neighbor matching algorithm and considering sex and age classes (5-year intervals) as matching covariates.
Sampling Method: Probability Sample
Enrollment: 608 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
QALY | baseline and 2 years
  quality-adjusted life-year. QALY scores range from 1 (perfect health) to 0 (dead)
DALY | baseline and 2 years
  Disability Adjusted Life Years. Disability-adjusted life years (DALYs) are a measure of overall disease burden, expressed as the number of years lost due to ill-health, disability, or early death.

CONTACTS AND LOCATIONS:
Locations (1):
- Local Health Authority of Taranto, Taranto, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: MISTRAL project — https://cordis.europa.eu/project/id/101095119/es